CLINICAL TRIAL: NCT04676594
Title: Validation of a Radiologic Tool for Diagnosing Pulmonary Fibrosis
Brief Title: Genentech Validation Tool for Pulmonary Fibrosis
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAS7955
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosis of Pulmonary Fibrosis on Chest CT: Retrospective chart review of patients with a diagnosis of pulmonary fibrosis on chest CT.

SUMMARY:
Radiology is an important component of the multidisciplinary team. The primary goal of this project will be to create a tool using findings on chest computed tomography (CT) for nearly 300 patients with the most common types of fibrosis. The tool will be tested using chest CT scans of an additional 100 patients with the 3 most common diagnoses of fibrosis. The second objective will be to further validate the tool by performing a reader study with 3 co-investigating radiologists and ask them to look at 100 CT scans of patients with fibrosis without tool and then with tool and see if accuracy of diagnosis improves compared to the working diagnosis when using the tool.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective review of adults (age > 21) with diagnosis of pulmonary fibrosis on chest CT and a pulmonologist report in electronic medical record confirming the working diagnosis from 1/1/2010 through 7/1/2019.

Exclusion Criteria:

* Failure to meet inclusion criteria including age < 21 and lack of a pulmonologists report in the medical record with a working diagnosis of patient's type of pulmonary fibrosis.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of usual interstitial pneumonitis, Chronic hypersensitivity pneumonitis or nonspecific interstitial pneumonitis and a chest CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Associations Between Patterns for CT Scan Features | Up to 6 months
  Creation of the radiologic diagnostic tool will be identified via statistical analysis of patterns for CT scan features. The patterns will be characterized using latent class analysis (LCA) and the demographic factors that are predictive of each pattern will be identified. Associations between patterns for CT scan features identified using LCA and the disease diagnosis will then be assessed using the Fisher's exact test.

SECONDARY OUTCOMES:
Cumulative Number of Accurate General Radiologist's Diagnoses of Fibrosis Type Without Diagnostic Tool | Up to 6 months
  The cumulative number of accurate (correct) diagnoses of fibrosis type (interstitial pneumonia (UIP), non-specific interstitial pneumonia (NSIP), or chronic hypersensitivity pneumonitis) without the diagnostic tool. Each assessment will be coded as correct or incorrect by comparing to the true disease diagnosis.
Cumulative Number of Accurate General Radiologist's Diagnoses of Fibrosis Type With Diagnostic Tool | Up to 6 months
  Cumulative number of accurate (correct) diagnoses of fibrosis type (interstitial pneumonia (UIP), non-specific interstitial pneumonia (NSIP), or chronic hypersensitivity pneumonitis) with the diagnostic tool. Each assessment will be coded as correct or incorrect by comparing to the true disease diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Salvatore, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No